CLINICAL TRIAL: NCT06936267
Title: Benefits of Early Proprioceptive Re-education Without Visual Information After Total Knee Arthroplasty
Acronym: RAPPEL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019/072/HP
Record Dates: First submitted 2025-04-04; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Unilateral Primary Osteoarthritis, Left Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proprioceptive exercise with eyes open (Active Comparator): * 30 minutes of techniques to increase joint amplitude
  * 15 to 30 minutes of muscular strengthening of the hamstrings against resistance (elastic or pulley), of the quadriceps without resistance and then against a light weight (1 to 2 kg).
  * 15 to 30 minutes of proprioceptive exercises, eyes open.
  * 10 to 15 minutes of functional exercises: walking, overcoming obstacles, going up and down stairs
  * 20 minutes of pressure therapy
  Interventions: Other: rehabilitation : eyes open
- proprioceptive exercise with eyes closed (Experimental): * 30 minutes of techniques to increase joint amplitude
  * 15 to 30 minutes of muscular strengthening of the hamstrings against resistance (elastic or pulley), of the quadriceps without resistance and then against a light weight (1 to 2 kg).
  * 15 to 30 minutes of proprioceptive exercises, eyes closed
  * 10 to 15 minutes of functional exercises: walking, overcoming obstacles, going up and down stairs
  * 20 minutes of pressure therapy
  Interventions: Other: rehabilitation : eyes closed

INTERVENTIONS:
Other: rehabilitation : eyes closed — proprioceptive exercise with eyes closed
  Arms: proprioceptive exercise with eyes closed
Other: rehabilitation : eyes open — proprioceptive exercise with eyes open
  Arms: proprioceptive exercise with eyes open

SUMMARY:
Osteoarthritis is a common and disabling joint disease, affecting 4.7% of men and 6.6% of women in France. It causes pain and impaired joint mobility, as well as a reduction in proprioception due to damage to intra-articular mechanoreceptors. In the long term, gonarthrosis can lead to limitations in activities of daily living and increase the risk of falls and institutionalisation.

Total knee arthroplasty is an effective treatment for reducing pain and improving functional capacity. However, 50% of patients operated on are not satisfied with the results obtained at 6 months, and between 37% and 55% experience no significant improvement in their functional mobility. It is therefore important to better define the modalities of rehabilitation interventions in order to improve their efficiency and the functional benefits for the patient.

Proprioception, the visual system and the vestibular system are the three major systems involved in posture and balance. Rehabilitation interventions aimed at improving balance involve these three inputs and their interaction. Studies have shown that proprioceptive rehabilitation can significantly improve balance and gait in patients who have undergone total knee arthroplasty. However, visual feedback may hinder the development of balance skills by limiting the use of other sensorimotor systems.

DETAILED DESCRIPTION:
The aim of this research project is to determine the benefits of visual deprivation and the methods of early proprioceptive exercises, right from the start of rehabilitation, on postural control in patients following total knee arthroplasty. Proprioceptive re-education with the eyes closed will be used from the very first rehabilitation sessions, evaluating its effect on proprioception. Currently, only one study has looked at the influence of the visual system in proprioceptive rehabilitation after total knee arthroplasty, seeking to assess the superiority of exercises with visual feedback compared with exercises without such feedback. The investigator presents an opposite and innovative questioning by proposing to evaluate on a larger scale the influence of visual deprivation rather than visual feedback.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 60 and 85 having undergone primary total knee arthroplasty for gonarthrosis
* Patient admitted to a Continuing Care and Rehabilitation (CCR) department and having received a maximum of 1 functional re-education session
* Patient able to remain in bipodal support with eyes closed for 30 seconds on inclusion
* Weight below the limit accepted by the posturography platform (100 kg)
* Patient having read and understood the information letter and having signed the consent form
* Affiliation with the social security system

Exclusion Criteria:

* Blindness
* Diabetes with peripheral neuropathy
* Central or peripheral nerve pathology (cerebellar syndrome, stroke sequelae, etc.)
* Previously known ataxia
* Alcoholism not withdrawn
* Pre-existing gait disorders making assessment impossible
* Disorders of the vestibular system
* Inflammatory rheumatism
* Length of stay in surgery > 7 days
* Person deprived of liberty by administrative or judicial decision or person placed under court protection / sub-guardianship or guardianship

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-06-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
the length of the projection of the centre of gravity on a posturography platform, in bipedal support, eyes closed, over 30 seconds | 3 weeks after randomization
  The main evaluation criterion is the length of the trace of the projection of the centre of gravity on a posturography platform, in bipedal support, eyes closed, over 30 seconds at 3 weeks (± 5 days) post-operatively or at discharge from the rehabilitation department, at the first intervening element.
  For this protocol, the posturographic analysis will be performed in the gait analysis laboratory of the Rouen Normandy University Hospital (Neurophysiology Department), by an investigator blinded to the treatment arm and trained in the use of the software.

CONTACTS AND LOCATIONS:
Overall Officials: Timothée GILLOT, Principal Investigator — UH ROUEN
Locations (2):
- France (2):
  - CRMPR - les herbiers, Bois-Guillaume
  - Chu Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No